CLINICAL TRIAL: NCT00273312
Title: An Open-label, Phase II Trial of Patupilone (EPO906) as Monotherapy to Evaluate Activity of Patupilone in Patients With Advanced Unresectable and/or Metastatic Hepatocellular Carcinoma (HCC)
Brief Title: Patupilone Activity in Advanced/Metastatic Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2213
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Advanced unresectable metastatic hepatocellular carcinoma; Liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — epothilone B

ARMS (1):
- Patupilone (Experimental): was administered at 10 mg/m2, as a single intravenous infusion over 20 minutes, once every 3 weeks
  Interventions: Drug: Patupilone

INTERVENTIONS:
Drug: Patupilone — Patupilone was in dosage strength of 10 mg/4 mL as a clear, colorless concentrate for solution for injection in individual 10 mL glass vials
  Other Names: EPO906

SUMMARY:
This study will evaluate the safety, efficacy, and activity of patupilone in patients with advanced unresectable and/or metastatic hepatocellular carcinoma based on tumor response using modified RECIST criteria.

ELIGIBILITY:
Inclusion criteria:

- Hepatocellular carcinoma patients with at least 1 previously un-irradiated, measurable lesion without any systemic single agent or combination chemotherapy. Previous local therapy is allowed.

Exclusion criteria:

Additional protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-01; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Tumor response as assessed by radiologic techniques and/or physical examination based on Response Evaluation Criteria in Solid Tumors (RECIST) | at screening and at completion of every 6 weeks prior to the next dose administration

SECONDARY OUTCOMES:
Time to progression | at screening and at completion of every 6 weeks prior to the next dose administration
Overall survival | at screening and at completion of every 6 weeks prior to the next dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Novartis Investigative Site, San Francisco, California, United States
- Hong Kong (2):
  - Novartis Investigative Site, Hong Kong, Shatin, NT
  - Novartis Investigative Site, Hong Kong
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Taiwan (2):
  - Novartis Investigative Site, Taipei, Taiwan ROC
  - Novartis Investigative Site, Tai Chung Municipality

REFERENCES:
- [Result] Zhou Q, Wong CH, Lau CP, Hui CW, Lui VW, Chan SL, Yeo W. Enhanced Antitumor Activity with Combining Effect of mTOR Inhibition and Microtubule Stabilization in Hepatocellular Carcinoma. Int J Hepatol. 2013;2013:103830. doi: 10.1155/2013/103830. Epub 2013 Feb 20. PMID 23509629